CLINICAL TRIAL: NCT04409496
Title: Chat-based Instant Messaging Support for Preventing Smoking Relapse in the Context of COVID-19 Outbreak: a Pilot Randomised Clinical Trial
Brief Title: Chat-based Support for Preventing Smoking Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tzu-Tsun Luk, Research Assistant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 20-356
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
Keywords: Instant messaging; Relapse prevention; WhatsApp; WeChat; Chat intervention; Chinese; Mobile health
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Chat-based instant messaging support + Self-help booklet
  Interventions: Behavioral: Chat-based instant messaging support; Behavioral: Self-help booklet
- Control group (Active Comparator): SMS message support + Self-help booklet
  Interventions: Behavioral: SMS message support; Behavioral: Self-help booklet

INTERVENTIONS:
Behavioral: Chat-based instant messaging support — Subjects will receive personalised instant messaging support for 12 weeks after baseline, address the five problems that contributed to smoking relapse:
  (1) lack of support for cessation, (2) negative mood or depression, (3) strong or prolonged withdrawal symptoms, (4) weight gain, and (5) smoking lapses. Updated information about the negative effect of smoking on risk of COVID-19 infection and prognosis will also be delivered.
  Arms: Intervention group
Behavioral: SMS message support — Subjects will receive regular SMS on generic smoking cessation for 3 months.
  Arms: Control group
Behavioral: Self-help booklet — Subjects will receive a standard self-help booklet on smoking relapse prevention.

SUMMARY:
This pilot trial aims to evaluate the effectiveness of chat-based instant messaging support in preventing smoking relapse in recent tobacco abstainers.

DETAILED DESCRIPTION:
Smoking cessation is one of the most cost-effective health interventions, which can add up to 10 years of life expectancy (Jha et al., 2013). However, it is very difficult to quit smoking because of the addictive effect of nicotine presents in tobacco products, and smokers typically make multiple attempts before successfully quit smoking. Providing evidence-based treatment could substantially increase the chance of successful quitting.

The Coronavirus Disease 2019 (COVID-19) provided new opportunities and challenges in promoting smoking cessation. A growing literature has shown that smoking is linked to poor progression of COVID-19 (Patanavanich & Glantz, 2020), which can be a new warning for motivating smokers to quit smoking. However, social distancing measures and increased stress and anxiety related to fear of contracting COVID-19 may increase the risk of smoking relapse in people who recently quit smoking (Patwardhan, 2020). There are also misinformation or unproven claims that smoking can protect against COVID-19. The social distancing measures also become a barrier for smokers who are interested in quitting to receive treatment from smoking cessation clinics. Therefore, implementing new interventions that can address the challenges in the context of the COVID-19 pandemic is needed.

Advance in mobile technologies provides a new avenue for delivering smoking cessation support. A qualitative interview of 21 current smokers in Hong Kong has found that mobile instant messaging app (e.g., WhatsApp) is an acceptable and feasible platform for providing chat support for smoking cessation (Luk et al., 2019). Chat-based support allows a registered nurse or trained counsellor to interact with a smoker individually through mobile instant messaging apps (e.g., WhatsApp and WeChat) and provide real-time, continuous, and personalized smoking cessation information and advice. A randomised trial of 1185 smokers found that the chat-based intervention integrated with brief intervention was effective in increasing smoking cessation (Wang et al., 2019). The trial also provided initial evidence that the intervention can be delivered as a stand-alone treatment or in combination with use of existing cessation treatment, to increase the chance of successful quitting. This study aims to adapt the chat intervention for smoking relapse prevention and evaluate its feasibility and effectiveness in recent tobacco abstainers enrolled in a clinic-based smoking cessation service in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 years or older
* Enrolled in a smoking cessation programme under Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation
* Daily tobacco use before service intake
* Not using any tobacco product for 3 to 30 days
* Own a mobile phone with a mobile instant messaging app (WhatsApp or WeChat) installed
* Able to communicate in Chinese (Cantonese or Mandarin)

Exclusion Criteria:

* Subjects with communication barriers owing to physical or cognitive conditions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Biochemically-validated tobacco abstinence | Assessed at 6 months after randomisation
  Defined by an exhaled carbon monoxide level of 3 parts per million or below

SECONDARY OUTCOMES:
Self-reported 6-month prolonged tobacco abstinence | Assessed at 6 months after randomisation
  Not more than five lapses permitted for 6 months after baseline
Self-reported 7-day point-prevalence tobacco abstinence | Assessed at 3 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 7-day point-prevalence tobacco abstinence | Assessed at 6 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported relapse rate | Assessed at 3 months after randomisation
  Defined as use of tobacco products for 7 consecutive days or longer
Self-reported relapse rate | Assessed at 6 months after randomisation
  Defined as use of tobacco products for 7 consecutive days or longer

OTHER OUTCOMES:
Change in self-efficacy to quit smoking | Assessed at 3 months after randomisation
  Assessed by the Chinese version of the Smoking Self-efficacy Questionnaire (SEQ-12), which contains 12 Likert items ranging from 1 (not certain at all) to 5 (very certain) with higher scores indicating greater perceived confidence in resisting smoking.
Change in self-efficacy to quit smoking | Assessed at 6 months after randomisation
  Assessed by the Chinese version of the Smoking Self-efficacy Questionnaire (SEQ-12), which contains 12 Likert items ranging from 1 (not certain at all) to 5 (very certain) with higher scores indicating greater perceived confidence in resisting smoking.
Nicotine withdrawal | Assessed at 3 months after randomisation
  Assessed by the Chinese verion of the Minnesota Nicotine Withdrawal Scale (MNWS), which contains 9 Likert items ranging from 0 (not at all) to 4 (very severe) with higher scores indicating greater nicotine withdrawal.
Nicotine withdrawal | Assessed at 6 months after randomisation
  Assessed by the Chinese verion of the Minnesota Nicotine Withdrawal Scale (MNWS), which contains 9 Likert items ranging from 0 (not at all) to 4 (very severe) with higher scores indicating greater nicotine withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Background] Patanavanich R, Glantz SA. Smoking Is Associated With COVID-19 Progression: A Meta-analysis. Nicotine Tob Res. 2020 Aug 24;22(9):1653-1656. doi: 10.1093/ntr/ntaa082. PMID 32399563
- [Background] Patwardhan P. COVID-19: Risk of increase in smoking rates among England's 6 million smokers and relapse among England's 11 million ex-smokers. BJGP Open. 2020 Jun 23;4(2):bjgpopen20X101067. doi: 10.3399/bjgpopen20X101067. Print 2020. No abstract available. PMID 32265183
- [Background] Luk TT, Wong SW, Lee JJ, Chan SS, Lam TH, Wang MP. Exploring Community Smokers' Perspectives for Developing a Chat-Based Smoking Cessation Intervention Delivered Through Mobile Instant Messaging: Qualitative Study. JMIR Mhealth Uhealth. 2019 Jan 31;7(1):e11954. doi: 10.2196/11954. PMID 30702431
- [Background] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Derived] Luk TT, Cheung YTD, Chan HC, Fok PW, Ho KS, Sze CD, Lam TH, Wang MP. Mobile Chat Messaging for Preventing Smoking Relapse Amid the COVID-19 Pandemic: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2023 Jan 5;25(2):291-297. doi: 10.1093/ntr/ntac045. PMID 35166327